CLINICAL TRIAL: NCT06506604
Title: "Psychological Intervention Enhanced by Virtual Reality for the Improvement of Appreciation of Body Functionality in Patients With Chronic Low-back-pain".
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Rosa M. Baños Rivera, Full Professor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PID2020-115609RB-C21
Record Dates: First submitted 2024-06-27; First posted 2024-07-17 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Chronic Low-back Pain

STUDY DESIGN:
Intervention Model Description: Multiple Baseline Single Case Design
Who Masked: Participant
Masking Description: Participants are blind to the variables of change.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Participants with low back pain. Multiple Base Line Single Case Design - 7 days wait (Experimental): Positive body image-based intervention. Main Components: Psychoeducation, Body Awareness, Acceptance, Functionality Appreciation and Gratitude toward the body.
  Interventions: Behavioral: CLEVER
- Participants with low back pain. Multiple Base Line Single Case Design - 10 days wait (Experimental): Positive body image-based intervention. Main Components: Psychoeducation, Body Awareness, Acceptance, Functionality Appreciation and Gratitude toward the body.
  Interventions: Behavioral: CLEVER
- Participants with low back pain. Multiple Base Line Single Case Design - 14 days wait (Experimental): Positive body image-based intervention. Main Components: Psychoeducation, Body Awareness, Acceptance, Functionality Appreciation and Gratitude toward the body.
  Interventions: Behavioral: CLEVER
- Participants with low back pain. Multiple Base Line Single Case Design - 11 days wait (Experimental): Positive body image-based intervention. Main Components: Psychoeducation, Body Awareness, Acceptance, Functionality Appreciation and Gratitude toward the body.
  Interventions: Behavioral: CLEVER

INTERVENTIONS:
Behavioral: CLEVER — CLEVER: A positive body image-based intervention for Chronic Low Back Pain.
  Patients will receive 4 sessions to approach 5 clinical modules: Pain Psychoeducation, Body Awareness, Pain Acceptance, Body Appreciation and Functionality and Gratitude. virtual reality environments will be used to enhance the clinical outcomes in two sessions. Each session will last 60 minutes.

SUMMARY:
The purpose of this study is to test whether a positive body image-based intervention is able to improve pain, disability, interference and emotional distress in people with chronic low back pain.

Patients will receive 4 sessions approaching 5 different clinical modules: Pain Psychoeducation, Body Awareness, Pain Acceptance, Body Appreciation and Functionality and Gratitude. 2 sessions will include virtual reality (VR) environments to enhance the clinical outcomes.

Researchers will analyse changes in the variables of interest after intervention compared to baseline.

DETAILED DESCRIPTION:
The purpose of this intervention is to examine the effects of a positive body image-based intervention using virtual reality to improve pain, interference and emotional distress.

The first session will be dedicated to psychoeducation about pain. Investigators will discuss what chronic pain is, what factors influence pain, chronification, body image and a brief presentation of the modules.

In the second session, a brief introduction to body awareness will be given and a VR environment will be used to carry out a body scan.

In the third session, Acceptance of pain will be worked on and a VR environment will be used to work on some variables related to the chronification of pain, such as paradoxical control or avoidance.

In the fourth session, the modules of Appreciation and Gratitude will be addressed.

Each session will last approximately one hour. First, participants will be screened to check eligibility inclusion/exclusion criteria. Second, eligible participants will complete baseline measures.

The study will be conducted following the principles stated in the Declaration of Helsinki.

The design chosen for the intervention will be a Multiple Baseline Single Case Design (SCD-MB). Data will be analysed by visual and statistical analysis. For visual analysis, the mean and/or median will be used to report the level, trend and stability of the 'within phase' data. For "between-phase" data, "Nonoverlap Statistics" such as "Nonoverlap of All Pairs" (NAP) will be used. For statistical analyses a Cohen's Difference of Means (Cohen's d) will be used to estimate the effect size at the individual level and multilevel analyses for across-case effect sizes.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with low back pain.

Exclusion Criteria:

* Meeting any of the following medical conditions:

  * Spinal tumor, infection or fracture
  * Systemic disease (autoimmune, infectious, vascular, endocrine, metabolic...)
  * Fibromyalgia
  * Cauda equina syndrome
  * History of spinal surgery
  * Musculoskeletal injury of lower extremities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2024-06-03 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Body Disability | The whole scale will be administered at the beginning (day 1 of 43) and the end of the intervention (day 43 of 43).
  Roland-Morris Questionnaire (RMQ) is a 24-item patient-reported outcome measure those inquiries about pain-related disability. Items are scored 0 if left blank or 1 if endorsed, for a total RMQ score ranging from 0 to 24.
Emotional Distress | The whole scale will be administered at the beginning (day 1 of 43) and the end of the intervention (day 43 of 43).
  The 4-item Brief Assessment of Distress about Pain (BADP) scale was developed to assess anxiety, fear, and depression related to pain, as well as an overall evaluation of distress about pain. Items are scored from 0 ("Not at all") to 4 ("Extreme"), for a total BADP score ranging from 0 to 16.
Pain Interference and Pain Intensity | The whole scale will be administered at the beginning (day 1 of 43) and the end of the intervention (day 43 of 43).
  The Brief Pain Inventory (BPI) scale was developed to assess the severity of pain and its impact on functioning. The scale consists of 9 items with qualitative and quantitative data on the following dimensions: "Worst pain in last 24 hours", "Least pain in last 24 hours", "Pain on average" and "Pain right now".
Level of Quality of Life | The whole scale will be administered at the beginning (day 1 of 43) and the end of the intervention (day 43 of 43).
  The EuroQol-5D (EQ-5D) scale is a 5-item scale to assess the quality of life of patients with several pathologies, chronic pain included. The individual assesses his or her own state of health, first in levels of severity by dimensions (descriptive system) and then on a more general visual analogue scale (VAS).

SECONDARY OUTCOMES:
Fear of movement | The whole scale will be administered at the beginning (day 1 of 43) and the end of the intervention (day 43 of 43).
  The Tampa Scale for Kinesophobia (TSK-11SV) is an 11-item scale that measures kinesophobia with statements asking the subject to answer from 1 ("Strongly disagree"), to 4 ("Strongly agree").
  Two items: 'I'M AFRAID OF UNINTENTIONALLY INJURING MYSELF', ´PHYSICAL ACTIVITY AGGRAVATES MY PAIN´ will be administered daily for 43 days via MPATH
Body Awareness | The whole scale will be administered at the beginning (day 1 of 43) and the end of the intervention (day 43 of 43) and one of the items of the scale: 'I NOTICE WHEN I FEEL UNCOMFORTABLE IN MY BODY´ will be administered daily for 43 days via MPATH.
  Dimensions of "Not Worrying" (items 9, 10 and 11), "Not distracting" (items 5, 6 and 7) and "Trusting" (items 30, 31 and 32) from the Multidimensional Assessment of Interoceptive Awareness (MAIA) will be used. This scale is a state-trait self-report questionnaire to measure multiple dimensions of interoception (awareness of bodily sensations). These dimensions have been chosen for their relationship to the intervention components and for their good psychometric quality. The scores range from 0 to 5, where higher scores indicate a higher level in that dimension.
Body Awareness | The whole scale will be administered at the beginning (day 1 of 43) and the end of the intervention (day 43 of 43).
  The following items have been created ad-hoc for this experiment:
  1. In general, I am able to pay attention to both pleasant and unpleasant bodily sensations.
  2. When I feel pain, I am also able to notice pleasant bodily sensations.
  3. Today I have noticed pleasant bodily sensations.
  4. Today I have noticed unpleasant bodily sensations.
  5. I am able to notice and differentiate the various sensations I experience in my body, regardless of whether they are pleasant or unpleasant (examples).
  6. I have the ability to pay attention to body signals, whether positive or negative.
  7. I am aware of physical sensations in my body, whether pleasant or uncomfortable.
  One of the items of the scale: 'TODAY I HAVE NOTICED PLEASANT BODILY SENSATIONS´ and 'TODAY I HAVE NOTICED UNPLEASANT BODILY SENSATIONS´ will be administered daily for 43 days via MPATH.
Chronic Pain Acceptance | The whole scale will be administered at the beginning (day 1 of 43) and the end of the intervention (day 43 of 43).
  Chronic Pain Acceptance Questionnaire 8 (CPAQ-8). Numerical rating scale ranging from 0 "Never true" to 6 "Always true" where higher scores indicate a higher Chronic Pain Acceptance (Pain Willingness and Activity Engagement).
  Two items: 'WHETHER I FELT PAIN OR NOT, I HAD A SATISFACTORY DAY´ and 'WHETHER I FELT PAIN OR NOT, I HAVE HAD A SATISFYING DAY TODAY´ will be administered daily for 43 days via MPATH.
Body Appreciation | The whole scale will be administered at the beginning (day 1 of 43) and the end of the intervention (day 43 of 43) and one of the items of the scale -'I FEEL LOVE AND RESPECT FOR MY BODY'- will be administered daily for 43 days via MPATH.
  Body Appreciation Scale 2 (BAS-2). Numerical rating scale ranging from 1 "Never" to 5 "Always", 10 items where higher scores indicate a higher Appreciation of the body.
Appreciation of Body Functionality | The whole scale will be administered at the beginning (day 1 of 43) and the end of the intervention (day 43 of 43).
  Functionality Appreciation Scale (FAS). The scores range from 1 to 5, where higher scores indicate higher levels of appreciation of body functionality.
  Two items of the scale -'I APPRECIATE MY BODY FOR WHAT IT IS ABLE TO DO'- and -'I AM GRATEFUL THAT MY BODY ALLOWS ME TO BE INVOLVED IN ACTIVITIES THAT I ENJOY OR THAT SEEM IMPORTANT TO ME´ will be administered daily for 43 days via MPATH
Pain Catastrophizing | The whole scale will be administered at the beginning (day 1 of 43) and the end of the intervention (day 43 of 43).
  The Pain Catastrophizing Scale (PCS) consists of 13 statements containing a number of thoughts and feelings typically present in the experience of pain. The items are divided into 3 categories: rumination, magnification and helplessness, with each item scored on a 5-point scale. The patient is asked to indicate the frequency with which these feelings or thoughts appear from 0 ("Not at all") to 4 ("All the time").
  Two of the items of the scale: -'I'M AFRAID THE PAIN WILL GET WORSE'- and -'I CAN'T STOP THINKING ABOUT HOW MUCH IT HURTS'- will be administered daily for 43 days via MPATH
Depression | The whole scale will be administered at the beginning (day 1 of 43) and the end of the intervention (day 43 of 43).
  The Patient Health Questionnaire (PHQ-9). The scale is composed of 9 items to assess depressive symptoms and the patient is asked to indicate the frequency with which these feelings, thoughts or states appear from 0 ("Not at all) to 3 ("Nearly every day").
Anxiety | The whole scale will be administered at the beginning (day 1 of 43) and the end of the intervention (day 43 of 43).
  The Generalised Anxiety Disorder-7 (GAD-7) scale is composed of 7 items to assess the different dimensions of the Generalised Anxiety Disorder and the patient is asked to mark the frequency from 'Never' to 'almost every day' in the last two weeks.

OTHER OUTCOMES:
Negative affect | This item will be administered daily for 43 days via MPATH
  How do you feel today? 0 = Not negative at all; 100 = Very negative
Positive affect | This item will be administered daily for 43 days via MPATH
  How do you feel today? 0 = Not positive at all; 100 = Very positive

CONTACTS AND LOCATIONS:
Overall Officials: Rosa M. Baños, PhD, Principal Investigator — University of Valencia
Locations (1):
- Arnau de Vilanova Hospital, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Valenzuela-Moguillansky C, Reyes-Reyes A, Gaete MI. Exteroceptive and Interoceptive Body-Self Awareness in Fibromyalgia Patients. Front Hum Neurosci. 2017 Mar 13;11:117. doi: 10.3389/fnhum.2017.00117. eCollection 2017. PMID 28348526
- [Background] Bailey KA, Gammage KL, van Ingen C, Ditor DS. "It's all about acceptance": A qualitative study exploring a model of positive body image for people with spinal cord injury. Body Image. 2015 Sep;15:24-34. doi: 10.1016/j.bodyim.2015.04.010. Epub 2015 May 21. PMID 26002149
- [Background] Alleva JM, Diedrichs PC, Halliwell E, Peters ML, Dures E, Stuijfzand BG, Rumsey N. More than my RA: A randomized trial investigating body image improvement among women with rheumatoid arthritis using a functionality-focused intervention program. J Consult Clin Psychol. 2018 Aug;86(8):666-676. doi: 10.1037/ccp0000317. PMID 30035583
- [Background] Kratochwill TR, Levin JR. Enhancing the scientific credibility of single-case intervention research: randomization to the rescue. Psychol Methods. 2010 Jun;15(2):124-44. doi: 10.1037/a0017736. PMID 20515235